CLINICAL TRIAL: NCT03639194
Title: A Phase I Study of ABBV-011 as a Single-Agent and in Combination With Budigalimab (ABBV-181) in Subjects With Relapsed or Refractory Small Cell Lung Cancer
Brief Title: A Study of ABBV-011 Alone and in Combination With Budigalimab (ABBV-181) in Participants With Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M17-327
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Cancer; Small Cell Lung Cancer; Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A: ABBV-011 Dose Escalation (Experimental): ABBV-011 via intravenous administration at various doses and dosing regimens until the maximum tolerated dose and/or the recommended Part B dose(s) is declared.
  Interventions: Drug: ABBV-011
- Part B: ABBV-011 Dose Expansion (Experimental): ABBV-011 via intravenous administration at dose regimen(s) that will not exceed the maximum tolerated dose determined in Part A.
  Interventions: Drug: ABBV-011
- Part C: ABBV-011 + Budigalimab Escalation and Expansion (Experimental): ABBV-011 via intravenous administration at various doses and dosing regimens starting at least 1 dose level below the recommended single-agent dose of ABBV-011 for Part B plus Budigalimab via intravenous administration at fixed doses and various dosing regimens.
  Interventions: Drug: ABBV-011; Drug: Budigalimab
- Part D: ABBV-011 Dose Evaluation for Japan (Experimental): ABBV-011 via intravenous administration will be administered every 3 weeks (Q3wk), on Day 1 of each 21-day cycle or alternate dosing regimens.
  Interventions: Drug: ABBV-011

INTERVENTIONS:
Drug: ABBV-011 — Intravenous
  Other Names: SC-011
Drug: Budigalimab — Intravenous
  Other Names: ABBV-181
  Arms: Part C: ABBV-011 + Budigalimab Escalation and Expansion

SUMMARY:
This is a multicenter, open-label, Phase 1 study of ABBV-011 given as a single agent and in combination with budigalimab (ABBV-181) in participants with relapsed or refractory small cell lung cancer (SCLC). The study consists of 4 parts: Part A is a single-agent ABBV-011 dose regimen finding cohort; followed by Part B, a single-agent ABBV-011 dose expansion cohort; and then Part C, an ABBV-011 and budigalimab (ABBV-181) combination escalation and expansion cohort; Part D, single-agent ABBV-011 dose-evaluating cohort for Japan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC) that is relapsed or refractory following at least 1 prior platinum-containing chemotherapy, but no more than 3 total prior lines of therapy, and with no curative therapy available.
* Measurable disease, defined as at least 1 tumor lesion greater than or equal to 10 mm in the longest diameter or a lymph node greater than or equal to 15 mm in short axis measurement assessed by computed tomography (CT) scan, according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Minimum life expectancy of at least 12 weeks.
* Recovery to at least Grade 1 of any clinically significant toxicity (excluding alopecia) prior to initiation of study drug administration.
* Adequate hematologic, hepatic, neurologic, and renal function.
* All participants in Part B and Part C will be required to have tumor tissue that tests positive for target expression.
* Sponsor may elect for confirmed SCLC tumor tissue to test positive for target expression for Parts A and D participants as well.
* Last dose of any prior anticancer therapy >= 4 weeks before the first dose of study drug.

Additional Inclusion Criteria for Study Part B and Part C:

* SCLC tumor tissue that tests positive for seizure-related homolog 6 (SEZ6) by immunohistochemistry (IHC).

Exclusion Criteria:

* History of confirmed or suspected liver cirrhosis, hepatic veno-occlusive disease (VOD), sinusoidal obstruction syndrome (SOS), alcohol dependence, or ongoing excessive alcohol use.
* Prior history of allogeneic or autologous stem cell transplantation.
* Documented history of stroke or clinically significant cardiac disease as described in the protocol within 6 months prior to the first dose of study drug.
* History of cardiac conduction abnormalities as described in the protocol.
* Recent or ongoing serious infection, as described in the protocol.
* Active SARS-CoV-2 infection.
* Prior or concomitant malignancies with some exceptions, as described in the protocol.
* Any significant medical or psychiatric condition, including any suggested by Screening laboratory findings, that in the opinion of the Investigator or Sponsor may place the participant at undue risk from the study treatment, interfere with interpretation of study results, or compromise ability to comply with protocol requirements.
* Participants with a history of hypersensitivity to the active ingredients or any excipients of study drugs (ABBV-011 or budigalimab [ABBV-181]) will be excluded.

Additional Exclusion Criteria for Part C:

* History of inflammatory bowel disease.
* Peripheral neuropathy Grade 2 with pain, or Grade 3 or higher.
* Body weight less than 35 kilograms.
* Active pneumonitis or interstitial lung disease (ILD) or a history of pneumonitis/ILD requiring treatment with steroids.
* Participants previously treated with an anti PD-1/PD-L1 targeting agent must meet additional criteria described in the protocol.
* Participant is judged by the Investigator to have evidence of ongoing hemolysis.
* Immunosuppressive use with exceptions as per protocol.
* Participants who have received a live vaccine within 30 days of start of study treatment.
* Active autoimmune disease with exceptions as indicated in the protocol.
* History of primary immunodeficiency, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
* Participants with a history of Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), or drug reaction with eosinophilia and systemic symptoms (DRESS).

Additional exclusion criteria for Japanese and Korean participants:

- Participants with a history of interstitial lung disease (pneumonitis) or current interstitial lung disease (pneumonitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to approximately 5 years after the first participant receives first dose of study drug
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RPTD) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  The Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RPTD) of ABBV-011 will be determined during the Part A dose escalation cohort.
Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RPTD) of ABBV-011 in Combination with Budigalimab | Up to approximately 5 years after the first participant receives first dose of study drug
  The Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RPTD) of ABBV-011 in combination with budigalimab will be determined during the Part C dose escalation cohort.
Number of Participants With Dose Limiting Toxicities (DLTs) | Up to approximately 5 years after the first participant receives first dose of study drug
  DLTs are adverse events as described in the protocol.
Mean Change from Baseline in Vital Signs | Up to approximately 5 years after the first participant receives first dose of study drug
  Mean change from Baseline in vital signs like blood pressure will be assessed.
Incidence of Laboratory Abnormaities | Up to approximately 5 years after the first participant receives first dose of study drug
  Number of participants with lab abnormalities will be assessed.
Mean Change from Baseline in Electrocardiogram (ECG) Parameters | Up to approximately 5 years after the first participant receives first dose of study drug
  Mean change from Baseline in ECG parameters like QTc interval will be assessed.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Maximum Serum Concentration (Cmax) of ABBV-011.
Area Under the Serum Concentration-Time Curve (AUCinf) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Area under the serum concentration-time curve within a dosing interval of ABBV-011.
Area Under the Serum Concentration-Time Curve within a Dosing Interval (AUC0-t) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Area under the serum concentration-time curve within a dosing interval (AUC0-t) of ABBV-011.
Time to Maximum Serum Concentration (Tmax) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Time to maximum serum concentration (Tmax) of ABBV-011.
Observed Serum Concentration at Trough (Ctrough) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Observed serum concentration at trough (Ctrough) of ABBV-011.
Apparent Terminal Half-Life (T1/2) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Apparent terminal half-life (T1/2) of ABBV-011.
Accumulation Ratio of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Accumulation ratio of ABBV-011.
Serum Clearance (CL) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Serum clearance of ABBV011.
Steady State Volume of Distribution (Vss) of ABBV-011 | Up to approximately 5 years after the first participant receives first dose of study drug
  Steady state volume of distribution (Vss) of ABBV-011.
Incidence of Antidrug Antibodies (ADA) Against ABBV-011 or Budigalimab (ABBV-181) | Up to approximately 5 years after the first participant receives first dose of study drug
  Number of participants with incidence of ADAs against ABBV-011 or budigalimab will be assessed.
Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to approximately 5 years after the first participant receives first dose of study drug
  ORR is defined as the percentage of participants with confirmed Complete Response (CR) or Partial Response (PR).
Clinical Benefit Rate (CBR) | Up to approximately 5 years after the first participant receives first dose of study drug
  CBR is defined as the percentage of participants with best overall response (confirmed or unconfirmed) of CR, PR or stable disease (SD).
Duration of Response (DOR) | Up to approximately 5 years after the first participant receives first dose of study drug
  DOR is defined as the time from the participant's initial objective response (CR or PR) to Progressive Disease (PD) or death due to any cause, whichever occurs first.
Duration of Clinical Benefit (DOCB) | Up to approximately 5 years after the first participant receives first dose of study drug
  (DOCB) is defined as the time from the participant's initial observation of clinical benefit (CR or PR or SD) to PD or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) | Up to approximately 5 years after the first participant receives first dose of study drug
  PFS time is defined as the time from the subject's first dose of study drug (Day 1) to either the subject's disease progression (PD) or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 5 years after the first participant receives first dose of study drug
  OS is defined as the time from the subject's first dose date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (32):
- United States (21):
  - University of Alabama at Birmingham - Main /ID# 207295, Birmingham, Alabama
  - Highlands Oncology Group, PA /ID# 207176, Springdale, Arkansas
  - University of California, Davis Comprehensive Cancer Center /ID# 207548, Sacramento, California
  - Yale School of Medicine /ID# 207559, New Haven, Connecticut
  - University of Iowa Hospitals and Clinics /ID# 207560, Iowa City, Iowa
  - University of Kentucky Chandler Medical Center /ID# 208217, Lexington, Kentucky
  - Massachusetts General Hospital /ID# 207549, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 213032, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center /ID# 207177, Ann Arbor, Michigan
  - Henry Ford Hospital /ID# 233539, Detroit, Michigan
  - Washington University-School of Medicine /ID# 207168, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 208216, New York, New York
  - Duke Cancer Center /ID# 207547, Durham, North Carolina
  - UH Cleveland Medical Center /ID# 207561, Cleveland, Ohio
  - The Ohio State University /ID# 207552, Columbus, Ohio
  - Tennessee Oncology, PLLC /ID# 207175, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center /ID# 207551, Nashville, Tennessee
  - NEXT Oncology /ID# 207167, San Antonio, Texas
  - University of Utah /ID# 207553, Salt Lake City, Utah
  - University of Washington /ID# 207557, Seattle, Washington
  - Univ of Wisconsin Hosp/Clinics /ID# 207556, Madison, Wisconsin
- Japan (5):
  - National Cancer Center Hospital East /ID# 230943, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center /ID# 229737, Matsuyama, Ehime
  - Hokkaido Cancer Center /ID# 229101, Sapporo, Hokkaido
  - Shizuoka Cancer Center /ID# 230911, Sunto-gun, Shizuoka
  - Wakayama Medical University Hospital /ID# 229111, Wakayama, Wakayama
- South Korea (5):
  - National Cancer Center /ID# 240169, Goyang, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 234274, Seongnam, Gyeonggido
  - Yonsei University Health System Severance Hospital /ID# 239515, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 234272, Seoul
  - Asan Medical Center /ID# 234273, Seoul
- National Cheng Kung University Hospital /ID# 234267, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiedemeyer WR, Gavrilyuk J, Schammel A, Zhao X, Sarvaiya H, Pysz M, Gu C, You M, Isse K, Sullivan T, French D, Lee C, Dang AT, Zhang Z, Aujay M, Bankovich AJ, Vitorino P. ABBV-011, A Novel, Calicheamicin-Based Antibody-Drug Conjugate, Targets SEZ6 to Eradicate Small Cell Lung Cancer Tumors. Mol Cancer Ther. 2022 Jun 1;21(6):986-998. doi: 10.1158/1535-7163.MCT-21-0851. PMID 35642431